CLINICAL TRIAL: NCT04415710
Title: Investigation of the Relationship Between the Pelvic Floor and Sexual Dysfunction in Women with Sjogren's Syndrome
Brief Title: Pelvic Floor and Sexual Dysfunction in Women with Sjogren's Syndrome
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, PhD Student, Akdeniz University
Other Study IDs: 2019-166
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2020-06

CONDITIONS: Sexual Dysfunction; Pelvic Floor Disorders; Pelvic Organ Prolapse; Urinary Incontinence; Constipation
Keywords: pelvic pain; sexual dysfunction; unirary incontinence; constipation; pelvic floor dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Pelvic Floor Disorders; Pelvic Organ Prolapse; Urinary Incontinence; Constipation; Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: Women with diagnosed Sjogren syndrome

SUMMARY:
Sjogren's syndrome (SS) is a chronic, systemic, autoimmune disease characterized by lymphocytic infiltration of all exocrine glands, especially tear and salivary glands, and is more common in women.

DETAILED DESCRIPTION:
Sexual functions are affected by symptoms such as pain, fatigue, stiffness, and hormonal imbalance in rheumatological disorders. Vaginal dryness and dyspepsia negatively affect participation in sexual activity. The aim of the study is to examine the pelvic floor problems of women with SS with a self-report, to compare them with healthy individuals, and finally to examine the relationship between pelvic floor problems and sexual dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18-65
* being a woman,
* having sex partner,
* no smoking, no alcohol

Exclusion Criteria:

* physical, psychological, cognitive impairment,
* having a non-Sjögren additional disease,
* malignancy,
* pregnancy,
* no urogenital disease,
* sarcoidosis,
* AIDS,
* anticholinergic drug use,
* had a gynecological or urological operation other than cesarean

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 94 women with Sjögren syndrome with an average age of 48.15 ± 8.73 years were included in the study. 94 women diagnosed as SS according to 2016 ACR-EULAR Classification Criteria for primary Sjögren's syndrome were included in the study by Rheumatology Clinic of Hospital. Ethical approval of the study was obtained from the Interventional Clinical Research Ethics Committee. All women were informed verbally and informed consent forms were signed.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Distress Inventory PFDI-20 | 1 week
  Pelvic Floor Distress Inventory has a total of 20 questions and 3 scales (Urinary Distress Inventory, Pelvic Organ Prolapse Distress Inventory, and Colorectal-Anal Distress Inventory). Each short-form scale demonstrates significant correlation with their long-form scales
Pelvic Floor Impact Questionnaire PFIQ | 1 week
  Pelvic Floor Impact Questionnaire (PFIQ): The questionnaire has 7 questions and each question has 3 separate responses. The response to each item of satisfaction, impact and worry was rated from 3 (quite a bit) to 0 (not at all) for the PFIQ-7. The mean value for all the answered items within the corresponding scale (possible value 0-3) was estimated, then multiplied by (100/3) to obtain the scale score, range 0-100.
Female Sexual Dysfunction Index FSFI | 1 week
  The FSFI is a brief questionnaire measure of sexual functioning in women. It was developed for the specific purpose of assessing domains of sexual functioning (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Ayan, Study Director — University of Health Sciences Antalya Training and Research Hospital
Locations (1):
- Ayse Ayan, Antalya, Turkey, Turkey (Türkiye)

REFERENCES:
- [Background] Budden AK, Te West NI, Sturgess AD, Moore KH. Pelvic floor dysfunction in female Sjogren's syndrome: an 8-year audit. Int Urogynecol J. 2016 Sep;27(9):1367-73. doi: 10.1007/s00192-016-2985-9. Epub 2016 Mar 10. PMID 26965411
- [Background] van Nimwegen JF, Arends S, van Zuiden GS, Vissink A, Kroese FG, Bootsma H. The impact of primary Sjogren's syndrome on female sexual function. Rheumatology (Oxford). 2015 Jul;54(7):1286-93. doi: 10.1093/rheumatology/keu522. Epub 2015 Feb 4. PMID 25652072